CLINICAL TRIAL: NCT06564649
Title: A Pilot Clinical Trial to Evaluate the Feasibility and Acceptability of: A Prospective, Unblinded, Randomized-controlled, Multicenter Biomarker Intervention Trial of a Urinary CXCL10 Clinical Surveillance Program in Pediatric Kidney Transplant Recipients for Early Ascertainment and Treatment of Subclinical Allograft Inflammation and Preservation of Kidney Transplant Function
Brief Title: PROACT Pilot Trial
Status: Active, not recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: University of Toronto (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, Tom Blydt-Hansen, Associate Professor, Department of Pediatrics, Faculty of Medicine, University of British Columbia, University of British Columbia
Other Study IDs: H23-00306
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Interventional Group: Participants in the intervention group will have urinary CXCL10 testing done on the Ella Platform up to every month for a 2 year follow up.
  Interventions: Diagnostic Test: CXCL10 Monitoring at clinical frequency
- Non-Interventional Group: Participants in the control group will have the standard of care urine test done via the clinical lab.

INTERVENTIONS:
Diagnostic Test: CXCL10 Monitoring at clinical frequency — The intervention is the implementation of real-time, serial urinary CXCL10 monitoring, with protocolized further clinical responses in the setting of elevated urinary CXCL10 levels.
  Groups: Interventional Group

SUMMARY:
Kidney transplantation is considered the best option to treat end-stage kidney disease, but the recipient's immune system may respond with rejection to the transplanted organ, leading to permanent kidney damage and failure.

The current standard for rejection monitoring in transplanted recipients is regular blood creatinine testing and kidney biopsies. Creatinine doesn't detect rejection until damages had occurred, causing some amount of kidney failure, and kidney biopsies are only done at set timepoints.

A new test called CXCL10 is shown to be more effective in detecting rejection from previous research and can be done as often as needed. Therefore, The investigators are doing this randomized trial to test CXCL10 as part of clinical care and to help design a larger national clinical trial in the future.

DETAILED DESCRIPTION:
Kidney transplant offers hope to thousands of people living with chronic kidney disease, but the average five-year-old who gets a kidney transplant should expect to need a second transplant before they reach adulthood. In adults, transplantation extends patient survival by 30-40 years compared to dialysis. In children, almost 30% lose the transplant within 5 years, with acute rejection as the most common cause. Despite the urgent need, approaches for monitoring and early acute rejection detection are largely unchanged for the past 20 years. The goal of this study is to introduce innovative monitoring that will permit timely acute rejection diagnosis and effective treatment, preserve kidney function, delay graft failure and spare the lives of children with chronic kidney failure.

In pediatric kidney transplants, a single episode of acute rejection confers up to a 19-fold increased risk of histologically visible scarring, the hallmark sign of progressive graft damage. Acute acute rejection is associated with subsequent development of anti-donor HLA antibodies, and chronic types of antibody-mediated and T cell-mediated acute rejection that are refractory to treatment. Acute rejection is readily treated with IV corticosteroids or depleting anti-thymocyte antibody treatments. These major adverse outcomes from acute rejection can only be mitigated or avoided if acute rejection is 1) identified and treated early before chronic inflammation is established; and 2) treated fully with confirmation that the acute inflammation has resolved.

The reported adverse outcomes relate predominantly to "clinical" presentations of acute rejection, i.e. those cases presenting with already worsening kidney failure. Subclinical acute rejection refers to the earlier phase of acute rejection where inflammation is onset but has not yet led to clinical graft dysfunction. This matters enormously because although acute rejection may be invisible to standard clinical monitoring, early identification and treatment of subclinical acute rejection improves long-term function and allograft survival. Acute rejection is a process, not an event. It starts with acute inflammation, and in the absence of immediate treatment it initiates a cascade of immune cytokine signals that causes memory types of effector cells to mature and leads to the suppression of regulatory types of immune cells that would otherwise promote tolerance to the allograft. This immune cell profile within the kidney is characteristic of chronic rejection and often co-exists in late-detected episodes of acute rejection.

Subclinical acute rejection is typically NOT associated with concurrent chronic inflammation or the presence of donor specific antibodies. With timely treatment of acute rejection, there is better preservation of histology, kidney function and survival . The pivotal trial by Rush et al., demonstrated that treatment of subclinical acute rejection detected by protocol surveillance biopsies improved long term outcome compared to clinical acute rejection monitoring and treatment. Natural history studies in adults and in children confirm the progressive nature of untreated subclinical acute rejection and the superior outcome when it is treated. Whether clinically detected or detected on biopsy surveillance (subclinical), both are considered as "acute rejection" and are treated similarly, based on the histological severity.

Unfortunately, damage related to delayed diagnosis and treatment is compounded by the lack of tools to evaluate treatment response. Although it is not standard, follow-up biopsies after acute rejection treatment reveal that 50-61% of children have persistent acute rejection subclinical 6-8 weeks after treatment - undetected by kidney function monitoring . Earlier diagnosis and treatment are therefore critical to prevent damage and preserve long-term function, as are interventions to ensure that reversal of subclinical inflammation is complete.

Acute rejection is much more common in children than in adults. This risk is compounded by the greater inefficacy of standard kidney function monitoring used for adults (serum creatinine) making it even harder to detect acute rejection in children or to monitor recovery after acute rejection treatment. This has led to a greater reliance on invasive kidney biopsies in children to surveil for subclinical acute rejection. Rates of surveillance biopsy-confirmed subclinical acute rejection reported in children range from 44-58% in the first year after transplant, much higher than in adults (4.2%).

Late acute rejection (>1 year post-transplant) in adolescence has an even worse prognosis, due to the extended periods of time with indolent and progressive inflammation before kidney failure is detected. Late acute rejection is beyond the post-transplant phase where routine biopsy surveillance is practical. This more entrenched and refractory inflammation is associated with 2 to 10-fold higher risk of chronic damage and graft failure compared to acute rejection in the first post-transplant year. Risk factors include non-adherence, which is also notoriously difficult to detect. Non-adherence is associated with higher rates late acute and chronic rejection, and is directly implicated in more than a third of pediatric renal allograft losses. Additional age-related and sex-related immune changes that peak in adolescence place this group at particularly high-risk. Timely detection of subclinical late acute rejection is currently impossible, since diagnosis requires already progressive functional deterioration to indicate a biopsy. Early acute rejection detection with new non-invasive tools could dramatically improve the outlook in these high-risk young people.

The investigators currently lack a reliable, noninvasive clinical test for subclinical acute rejection, which means that acute rejection may fester undetected until substantial kidney damage has occurred. The introduction of surveillance biopsies has led to earlier detection of subclinical acute rejection, improved allograft function and increased survival. However, concerns about procedure morbidity and cost have hindered widespread adoption of surveillance biopsies, in use at only 34% of pediatric transplant centers. These same issues practically limit their use for serial monitoring, especially after the first transplant year, highlighting the need for a noninvasive alternative.

There is ample evidence that urinary CXCL10 testing is very effective at both identifying acute rejection AND confirming response to treatment. Since 2004, there have been 19 reports that support its use for detection of subclinical acute rejection, including 4 reports in children. Other cytokines that have not been fully validated in children include CXCL9 and IL-6. Levels of urinary CXCL10 increase in advance of clinical acute rejection diagnosis and decreases after its treatment and resolution . Urinary CXCL10 is also effective at identifying inflammation from other important causes of graft injury, such as CMV interstitial nephritis, subclinical pyelonephritis and BK polyomavirus nephritis. Persistent elevation of urinary CXCL10 signals unresolved acute inflammation, such as from untreated or persistent subclinical acute rejection and is associated with chronic scarring and progressive kidney failure. Despite the wealth of evidence in support, CXCL10 testing has not yet been translated into routine practice because of the lack of studies that demonstrate clinical effectiveness to improve outcome.

This proposal will test the feasibility of a definitive clinical trial in transplanted children. The goal of the definitive clinical trial is to determine whether serial urinary CXCL10 monitoring will reduce the incidence of and severity of allograft failure. It will be a prospective, multicenter, randomized, controlled trial where the intervention is serial urinary monitoring of CXCL10 alongside routine clinical testing at 1-3-month intervals, with test results used to guide subsequent care decisions. Patients randomized to control will have standard of care monitoring, with biobanking of urine samples for later analysis. The primary outcome will be the difference in relative decline (from baseline) of kidney function after 2 years of monitoring. The will also collect preliminary data on validity of cytokines CXCL9 and IL-6, for potential inclusion in the definitive study.

This pilot study design is a prospective, multicenter, randomized, controlled study of the feasibility and acceptability of a definitive clinical trial. It will follow the same procedures as the definitive trial; however, the primary aims will be to demonstrate that logistical and recruitment requirements can be met as well as to collect economic data to inform the optimal testing procedure (local vs. central). The pilot will enroll 60 prevalent kidney transplant recipients who are >6 months post-transplant.

The objectives of this pilot trial are to evaluate the feasibility of a definitive trial:

1. Demonstrate capacity to recruit, randomize and retain 60 participants
2. Identify and resolve challenges in executing the study protocol regarding sample acquisition, CXCL10 testing, and adherence to the mandated trial protocols
3. Comparison of cost and logistical supports needed for local vs. central CXCL10 testing options

ELIGIBILITY:
Inclusion Criteria:

* Prevalent pediatric kidney transplant recipients (<19 years at transplantation) who are more than 6 months after transplant, with informed consent and assent.
* Must be available to follow-up for two years after initiation of urinary CXCL10 monitoring

Exclusion Criteria:

* Expected transfer to adult care in the next 2 years.
* In center routine follow-up interval >3 months between visits
* Non-adherence to routine transplant clinic visits.
* Recent acute rejection episode in the last 3 months prior to enrolment. Patients may be enrolled if rejection was more than 3 months prior to enrolment. No exclusion for donor-specific antibody in the absence of acute cellular or antibody-mediated rejection.
* Estimated glomerular filtration rate <30 ml/min/1.73m2 (stage IV/V CKD).
* Inability to reliably obtain urinary samples for monitoring purposes.
* Contraindication to kidney biopsy.

Ages: 6 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study includes prevalent pediatric kidney transplant recipients who are below 19 years of page at the time of transplant and who are more than 6 months after their transplant.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Capacity of Recruitment for future definitive trial | 8 months
  Demonstrate capacity to recruit, randomize and retain 60 participants

SECONDARY OUTCOMES:
Study Protocol Feasibility | 2 years
  2) Identify and resolve challenges in executing the study protocol regarding sample acquisition, CXCL10 testing, and adherence to the mandated trial protocols
Trial Cost and logistical support evaluation | 2 years
  3) Comparison of cost and logistical supports needed for local vs. central CXCL10 testing options

CONTACTS AND LOCATIONS:
Overall Officials: Tom BLydt-Hansen, MDCM, FRCPC, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - BC Children's Hospital, Vancouver, British Columbia
  - The Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data and results will be retained for use in the definitive clinical trial that is anticipated to follow the pilot trial. They may be further shared with any qualified investigator upon request, with approval of the principal investigator. The purpose of the data retention is to make data/samples available for ancillary studies related to the primary study, in collaboration with the PI after the primary study is complete.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Deidentified participant data will be retained for at least 5 years after primary study reporting to the sponsor has been completed.
Access Criteria: * Relevant Research Ethics Board Approval
  * Approval from the principal investigator

REFERENCES:
- [Background] Chua A, Cramer C, Moudgil A, Martz K, Smith J, Blydt-Hansen T, Neu A, Dharnidharka VR; NAPRTCS investigators. Kidney transplant practice patterns and outcome benchmarks over 30 years: The 2018 report of the NAPRTCS. Pediatr Transplant. 2019 Dec;23(8):e13597. doi: 10.1111/petr.13597. Epub 2019 Oct 27. PMID 31657095
- [Background] Smith JM, Martz K, Blydt-Hansen TD. Pediatric kidney transplant practice patterns and outcome benchmarks, 1987-2010: a report of the North American Pediatric Renal Trials and Collaborative Studies. Pediatr Transplant. 2013 Mar;17(2):149-57. doi: 10.1111/petr.12034. Epub 2013 Jan 2. PMID 23281637
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Karpinski M, Ho J, Storsley LJ, Goldberg A, Birk PE, Rush DN, Nickerson PW. Evolution and clinical pathologic correlations of de novo donor-specific HLA antibody post kidney transplant. Am J Transplant. 2012 May;12(5):1157-67. doi: 10.1111/j.1600-6143.2012.04013.x. Epub 2012 Mar 19. PMID 22429309
- [Background] Dart AB, Schall A, Gibson IW, Blydt-Hansen TD, Birk PE. Patterns of chronic injury in pediatric renal allografts. Transplantation. 2010 Feb 15;89(3):334-40. doi: 10.1097/TP.0b013e3181bc5e49. PMID 20145525
- [Background] Blydt-Hansen TD, Sharma A, Gibson IW, Mandal R, Wishart DS. Urinary metabolomics for noninvasive detection of borderline and acute T cell-mediated rejection in children after kidney transplantation. Am J Transplant. 2014 Oct;14(10):2339-49. doi: 10.1111/ajt.12837. Epub 2014 Aug 19. PMID 25138024
- [Background] Birk PE, Stannard KM, Konrad HB, Blydt-Hansen TD, Ogborn MR, Cheang MS, Gartner JG, Gibson IW. Surveillance biopsies are superior to functional studies for the diagnosis of acute and chronic renal allograft pathology in children. Pediatr Transplant. 2004 Feb;8(1):29-38. doi: 10.1046/j.1397-3142.2003.00122.x. PMID 15009838
- [Background] Landsberg A, Riazy M, Blydt-Hansen TD. Yield and utility of surveillance kidney biopsies in pediatric kidney transplant recipients at various time points post-transplant. Pediatr Transplant. 2021 Mar;25(2):e13869. doi: 10.1111/petr.13869. Epub 2020 Oct 19. PMID 33073499
- [Background] Blydt-Hansen TD, Gibson IW, Gao A, Dufault B, Ho J. Elevated urinary CXCL10-to-creatinine ratio is associated with subclinical and clinical rejection in pediatric renal transplantation. Transplantation. 2015 Apr;99(4):797-804. doi: 10.1097/TP.0000000000000419. PMID 25222013
- [Background] Blydt-Hansen TD, Sharma A, Gibson IW, Wiebe C, Sharma AP, Langlois V, Teoh CW, Rush D, Nickerson P, Wishart D, Ho J. Validity and utility of urinary CXCL10/Cr immune monitoring in pediatric kidney transplant recipients. Am J Transplant. 2021 Apr;21(4):1545-1555. doi: 10.1111/ajt.16336. Epub 2020 Oct 30. PMID 33034126
- [Background] Birk PE, Blydt-Hansen TD, Dart AB, Kaita LM, Proulx C, Taylor G. Low incidence of adverse events in outpatient pediatric renal allograft biopsies. Pediatr Transplant. 2007 Mar;11(2):196-200. doi: 10.1111/j.1399-3046.2006.00659.x. PMID 17300500
- [Background] Lamarche C, Sharma AK, Goldberg A, Wang L, Blydt-Hansen TD. Biomarker implementation: Evaluation of the decision-making impact of CXCL10 testing in a pediatric cohort. Pediatr Transplant. 2021 May;25(3):e13908. doi: 10.1111/petr.13908. Epub 2020 Nov 6. PMID 33155737
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Pochinco D, Birk PE, Ho J, Karpinski M, Goldberg A, Storsley L, Rush DN, Nickerson PW. Rates and determinants of progression to graft failure in kidney allograft recipients with de novo donor-specific antibody. Am J Transplant. 2015 Nov;15(11):2921-30. doi: 10.1111/ajt.13347. Epub 2015 Jun 10. PMID 26096305